CLINICAL TRIAL: NCT04454749
Title: Endometrial Compaction and Its Influence on Pregnancy Rate in Frozen Embryo Cycle Regimes
Status: Terminated | Type: Observational
Why Stopped: Investigators perogative
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Principal Investigator, Barbara Lawrenz, Scientific Director, ART Fertility Clinics LLC
Other Study IDs: 2003-ABU-002-BL
Record Dates: First submitted 2020-06-28; First posted 2020-07-01 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Endometrial Disorder; Infertility, Female; IVF; Pregnancy Early
Keywords: infertilty; progesterone; endometrium; pregnancy
MeSH Terms: conditions — Infertility, Female | interventions — Hematologic Tests; Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Stimulated cycles: Ovarian stimulation will be performed by standard protocols. Stimulation medication dosage will be individualised prior to stimulation start according to the ovarian reserve parameters and during ovarian stimulation according to the ovarian response and the measured levels of E2 and progesterone (P4), in order to avoid progesterone elevation during late follicular phase. Final oocyte maturation will be achieved by administration of either 10.000 IU of hCG, 0.3 mg of GnRH agonist (Triptorelin) or dual trigger (hCG and GnRH-analogue), as soon as ≥ 3 follicles ≥ 17 mm are present. Oocyte retrieval will be carried out 36 hours after administration of the trigger. Embryos will undergo PGT-A at blastocyst stage and be vitrified thereafter.
  Interventions: Diagnostic Test: Blood test; Diagnostic Test: Ultrasound
- Artificial (HRT) Cycles: Start of estradiol valerate 4mg on day 2 of the cycle for three days. Increase E2 to 6mg on day 4 of E2 treatment. E2 dose may be increased according to clinician discretion based on endometrial thickness. Maximum time of E2 exposure will be 14 days. Transvaginally scan to monitor endometrial development and to exclude the presence of a dominant follicle. Serial measurements of serum LH, estradiol and progesterone levels. Commence the initial progesterone dose of 100mg at 22hrs (vaginal suppository) after ≥ 7 days and ≤ 16 days of estradiol administration when the minimal endometrial thickness achieved is 6mm with a trilaminar appearance. Subsequently increase progesterone administration to 100mg vaginally three times daily. Continue estradiol administration 6mg (3 tablets daily).
  Blastocyst transfer is scheduled on the 5th full day of progesterone administration, following the initial initiation of progesterone.
  Interventions: Diagnostic Test: Blood test; Diagnostic Test: Ultrasound
- Spontaneous natural cycles: Ultrasound scans to monitor follicular growth and serial measurements of serum LH, estradiol and progesterone levels to determine the timing of ovulation. The LH surge will be considered to have begun when the concentration rises by 180% above the most recent serum value and continues to rise thereafter.
  Day 1 after the LH rise, a decrease in estradiol concentration is identified. Twenty four hours later progesterone concentrations rise with a level of greater than or equal to 1.5ng/ml confirming ovulation (day 0). This is considered as day 0 with initiation of vaginal progesterone 100mg (vaginal suppository) at 2200H. The following day (day 1) increases progesterone administration to 100mg vaginally three times daily (8 hourly) and continues this regime until 7 weeks gestation as per clinic protocol.
  Embryo transfer is scheduled 5 days (day 5) following confirmation of ovulation (day 0).
  Interventions: Diagnostic Test: Blood test; Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: Blood test — Mesurement of E2, P4, LH, FSH hormones
Diagnostic Test: Ultrasound — Follicular measurement and endometrium measurement

SUMMARY:
For a pregnancy to occur, an euploid embryo at blastocyst developmental stage, a receptive endometrium and the synchrony of both is crucial. Many studies lately investigated the influence of the endometrial thickness and pattern on the artificial reproductive technology (ART) outcome, however, with conflicting results.

DETAILED DESCRIPTION:
Further on, the measurement of the endometrial thickness was mostly performed either on the day of final oocyte maturation in stimulated cycles with fresh embryo transfer or on the day of progesterone administration in FET cycles.

Progesterone is essential for the secretory transformation and compaction of the endometrium, prior to implantation. A recently published paper (Haas et al., 2019) however, evaluated the degree of endometrial compaction under the influence of progesterone in FET cycles and described, that a lack of certain endometrial compaction has a negative impact on the ongoing pregnancy rate. As in this study embryos of unknown ploidy status were transferred, the role of embryo ploidy on the outcome may bias the study results.

In the herein presented study protocol we aim to investigate the influence of endometrial compaction in FET cycles in which euploid embryos are transferred.

HYPOTHESIS: Lack of endometrial compaction after the start of progesterone leads to an impaired reproductive outcome.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years to 40 years with regular menses (26-34 days)
* Having 1 or 2 chromosomally normal cryopreserved blastocysts available for transfer after IVF / ICSI treatment
* First frozen-thawed transfer cycle
* Progesterone level < 1.5 ng/mL day of trigger injection in stimulation cycle from which embryos to be transferred were created.

Exclusion Criteria:

* Polycystic ovarian syndrome
* Poor ovarian responder in accordance with Bologna criteria
* Uterine abnormality US / saline infusion sonohysterogram
* Previous dilatation & curettage (D&C)
* Hydrosalpinx
* Asherman syndrome
* History of endometriosis AFS ≥ 2
* ICSI due to severe male factor with testicular sperm
* Any known contraindications or allergy to oral estradiol or progesterone.
* Discontinuation of HRT medication ( medication error in research HRT cycle )
* Failure to detect ovulation in the research natural cycle
* Ovulation after day 20 in a natural cycle
* Duration of estradiol exposure ≥ 17 days and endometrium < 6mm
* Spontaneous ovulation in HRT artificial cycle

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Patients who are undergoing ovarian stimulation for IVF/ICSI with pre-implantation genetic screening and embryo vitrification, who are planned for their first FET transfer cycle.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 12 weeks
  Ongoing pregnancy rate (≥ 12 weeks) in patients with endometrial compaction compared to patients without endometrial compaction after frozen embryo transfer of 1 or 2 euploid blastocysts

SECONDARY OUTCOMES:
Biochemical pregnancy rate in HRT cycle | 5 weeks
  Positive hCG, but at 5 gestational weeks no ultrasonographic visible gestational sac seen after embryo transfer in HRT-FET cycles with one or two euploid embryos, depending on the degree of compaction.
Biochemical pregnancy rate in spontaneous cycle | 5 weeks
  positive hCG, but at 5 gestational weeks no ultrasonographic visible gestational sac seen) after embryo transfer in NC-FET cycles with one or two euploid embryos, depending on the degree of compaction.
Clinical implantation rate in HRT cycle | 6 weeks
  Number of gestational sacs observed by ultrasound at 6 weeks of gestation divided by the number of embryos transferred), defined by a ß-hCG of > 5 IU on day 12 after embryo transfer in HRT-FET cycles with one or two euploid embryos, depending on the degree of compaction
Clinical implantation rate in spontaneous cycle | 6 weeks
  Number of gestational sacs observed by ultrasound at 6 weeks of gestation divided by the number of embryos transferred), defined by a ß-hCG of > 5 IU on day 12 after embryo transfer in NC-FET cycles with one or two euploid embryos, depending on the degree of compaction.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Lawrenz, PhD, Principal Investigator — IVI Middle East Fertility Clinic LLC
Locations (1):
- IVI Middle East Fertility Clinic, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bu Z, Sun Y. The Impact of Endometrial Thickness on the Day of Human Chorionic Gonadotrophin (hCG) Administration on Ongoing Pregnancy Rate in Patients with Different Ovarian Response. PLoS One. 2015 Dec 30;10(12):e0145703. doi: 10.1371/journal.pone.0145703. eCollection 2015. PMID 26717148
- [Result] Fatemi HM, Kyrou D, Bourgain C, Van den Abbeel E, Griesinger G, Devroey P. Cryopreserved-thawed human embryo transfer: spontaneous natural cycle is superior to human chorionic gonadotropin-induced natural cycle. Fertil Steril. 2010 Nov;94(6):2054-8. doi: 10.1016/j.fertnstert.2009.11.036. Epub 2010 Jan 25. PMID 20097333
- [Result] Haas J, Smith R, Zilberberg E, Nayot D, Meriano J, Barzilay E, Casper RF. Endometrial compaction (decreased thickness) in response to progesterone results in optimal pregnancy outcome in frozen-thawed embryo transfers. Fertil Steril. 2019 Sep;112(3):503-509.e1. doi: 10.1016/j.fertnstert.2019.05.001. Epub 2019 Jun 24. PMID 31248618
- [Result] Irani M, Robles A, Gunnala V, Reichman D, Rosenwaks Z. Optimal parameters for determining the LH surge in natural cycle frozen-thawed embryo transfers. J Ovarian Res. 2017 Oct 16;10(1):70. doi: 10.1186/s13048-017-0367-7. PMID 29037231
- [Result] Kasius A, Smit JG, Torrance HL, Eijkemans MJ, Mol BW, Opmeer BC, Broekmans FJ. Endometrial thickness and pregnancy rates after IVF: a systematic review and meta-analysis. Hum Reprod Update. 2014 Jul-Aug;20(4):530-41. doi: 10.1093/humupd/dmu011. Epub 2014 Mar 23. PMID 24664156
- [Result] La Marca A, Sunkara SK. Individualization of controlled ovarian stimulation in IVF using ovarian reserve markers: from theory to practice. Hum Reprod Update. 2014 Jan-Feb;20(1):124-40. doi: 10.1093/humupd/dmt037. Epub 2013 Sep 29. PMID 24077980
- [Result] Lawrenz B, Labarta E, Fatemi H, Bosch E. Premature progesterone elevation: targets and rescue strategies. Fertil Steril. 2018 Apr;109(4):577-582. doi: 10.1016/j.fertnstert.2018.02.128. PMID 29653703
- [Result] Liu KE, Hartman M, Hartman A, Luo ZC, Mahutte N. The impact of a thin endometrial lining on fresh and frozen-thaw IVF outcomes: an analysis of over 40 000 embryo transfers. Hum Reprod. 2018 Oct 1;33(10):1883-1888. doi: 10.1093/humrep/dey281. PMID 30239738
- [Result] Liu Y, Ye XY, Chan C. The association between endometrial thickness and pregnancy outcome in gonadotropin-stimulated intrauterine insemination cycles. Reprod Biol Endocrinol. 2019 Jan 23;17(1):14. doi: 10.1186/s12958-019-0455-1. PMID 30674305
- [Result] Testart J, Frydman R, Feinstein MC, Thebault A, Roger M, Scholler R. Interpretation of plasma luteinizing hormone assay for the collection of mature oocytes from women: definition of a luteinizing hormone surge-initiating rise. Fertil Steril. 1981 Jul;36(1):50-4. doi: 10.1016/s0015-0282(16)45617-7. PMID 7250407
- [Result] Vaegter KK, Lakic TG, Olovsson M, Berglund L, Brodin T, Holte J. Which factors are most predictive for live birth after in vitro fertilization and intracytoplasmic sperm injection (IVF/ICSI) treatments? Analysis of 100 prospectively recorded variables in 8,400 IVF/ICSI single-embryo transfers. Fertil Steril. 2017 Mar;107(3):641-648.e2. doi: 10.1016/j.fertnstert.2016.12.005. Epub 2017 Jan 17. PMID 28108009
- [Result] Yuan X, Saravelos SH, Wang Q, Xu Y, Li TC, Zhou C. Endometrial thickness as a predictor of pregnancy outcomes in 10787 fresh IVF-ICSI cycles. Reprod Biomed Online. 2016 Aug;33(2):197-205. doi: 10.1016/j.rbmo.2016.05.002. Epub 2016 May 13. PMID 27238372
- [Result] Zhao J, Zhang Q, Wang Y, Li Y. Endometrial pattern, thickness and growth in predicting pregnancy outcome following 3319 IVF cycle. Reprod Biomed Online. 2014 Sep;29(3):291-8. doi: 10.1016/j.rbmo.2014.05.011. Epub 2014 Jun 13. PMID 25070912